CLINICAL TRIAL: NCT05231837
Title: Neighborhood Park Youth Sports Program Fee Waiver and Intensive Family Outreach to Promote Physical Activity in Low-Income Children Ages 6-12 Years
Brief Title: Neighborhood Park Youth Sports Program Fee Waiver and Intensive Family Outreach
Acronym: PARKS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00012450
Record Dates: First submitted 2022-01-29; First posted 2022-02-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Physical Activity
Keywords: Physical Activity Low Income Youth Parks
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Parks will be randomized to one of two conditions for a period of two years. Individual measures of physical activity and behavior will be collected among children and parents who reside in the neighborhoods that are served by each park. Children and parents will be enrolled for two years and measured at baseline, six, twelve and twenty-four months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fee Waiver (Experimental): Fees for youth sports programs will be waived in this condition. Youth who enroll in youth sports programs in parks that are randomly assigned to this condition will pay no fee for program enrollment.
  Interventions: Behavioral: Experimental: Fee Waiver
- Fee Waiver Plus Intensive Outreach (Experimental): Parks randomly assigned to the Intensive Outreach and Fee Waiver:
  Intensive Outreach consists of the formation and activity of a community advisory group who will engage with neighborhood community partners to support parents in the neighborhood to enroll their child and support the child's participation in the park youth sports programs offered at the neighborhood park and recreation center. Program marketing and materials and registration will be offered in both Spanish and English. Program coaches will be supported with technical assistance from study staff to implement the park youth sports program with high fidelity and with high communication and engagement with enrolled youth and their parents.
  Fees for youth sports programs will be waived in this condition. Youth who enroll in youth sports programs in parks that are randomly assigned to this condition will pay no fee for program enrollment.
  Interventions: Behavioral: Fee Waiver Plus Intensive Outreach

INTERVENTIONS:
Behavioral: Experimental: Fee Waiver — Fees are waived for youth sports programs at the park and recreation center
  Arms: Fee Waiver
Behavioral: Fee Waiver Plus Intensive Outreach — Fees are waived for youth sports programs at the park and recreation center and intensive outreach is conducted in the neighborhood through community advisory boards and partner engagement.
  Arms: Fee Waiver Plus Intensive Outreach

SUMMARY:
To evaluate a park-level intervention to increase child moderate/vigorous physical activity (MVPA), and decrease sedentary time among low-income racially/ethnically diverse children ages 6-12 yrs. Neighborhood parks (n=20) from Minneapolis (n=8) and Saint Paul (n=12) park systems will be randomized for a 2-year period to one of two arms: 1) Intensive Park Outreach and Youth Sports Program Fee Waiver (n=10); or 2) Youth Sports Program Fee Waiver Only (n=10). The evaluation cohort will consist of 432 children ages 6-12 yrs who reside in one of the 20 randomized park neighborhoods. Measurements from evaluation cohort-enrolled individual children will be collected at baseline, 6, 12, and 24 months.

DETAILED DESCRIPTION:
This research evaluates the effects of a park-level intervention to increase child moderate/vigorous physical activity (MVPA), and decrease sedentary time among low-income racially/ethnically diverse children ages 6-12 yrs. Neighborhood parks (n=20) from Minneapolis (n=8) and Saint Paul (n=12) park systems will be randomized for a 2-year period to one of two arms: 1) Intensive Park Outreach and Youth Sports Program Fee Waiver (n=10); or 2) Youth Sports Program Fee Waiver Only (n=10). In the Intensive Park Outreach and Youth Sports Program Fee Waiver condition, Community Advisory Boards (CABs) will be created to develop partner networks that will publicize the free youth park programs offered at the local park and recreation center. CABs will engage in program recruitment activities throughout the study to directly engage parents to support their child's PA through enrollment and participation in youth sports park programs. Parents will be supported through CAB outreach activities that address cultural and communication barriers, and financial barriers will be addressed through the fee waiver program. The Youth Sports Program Fee Waiver Only will consist of financial supports through the fee waiver, but will not include additional outreach beyond usual park outreach activities. The evaluation cohort will consist of 432 children ages 6-12 yrs who reside in one of the 20 randomized park neighborhoods. Measurements from evaluation cohort-enrolled individual children will be collected at baseline, 6, 12, and 24 months.

The Specific Aims of this research are:

Specific Aim 1: To evaluate the effects of a park-level intervention on changes in child MVPA over 6, 12 and 24 months.

Specific Aim 2: To evaluate the effects of a park-level intervention on changes in child sedentary behavior over 6, 12 and 24 months.

Exploratory Aim 3: To evaluate the effects of a park-level intervention on changes in parent light and sedentary activity over 6, 12 and 24 months.

Hypothesis 1: Children who live in a neighborhood where the park is randomized to intensive park outreach and fee waiver will have larger increases in MVPA and decreases in sedentary behavior at 6, 12 and 24 months relative to children who live in a fee waiver-only neighborhood.

Hypothesis 2: Parents of children who live in a neighborhood where the park is randomized to intensive park outreach and fee waiver will have larger increases in light PA and decreases in sedentary behavior at 6, 12, and 24 months relative to parents of children who live in a fee waiver-only neighborhood.

IMPACT: The proposed research will provide evidence about the effectiveness of a park-based intervention that includes intensive park outreach and youth sports program fee waivers on changes in physical activity among racially/ethnically diverse children with low-income. It will provide critical information needed to support policies and programs that increase the reach and participation of children living in high-risk, low income communities, and thereby reduce racial/ethnic and income-related physical activity disparities.

ELIGIBILITY:
Inclusion Criteria:

* age 6-12 years
* do not meet guidelines for recommended level of physical activity
* live in neighborhood served by one of 20 study parks
* able to be physically active
* do not plan to move in the next two years

Exclusion Criteria:

* younger than 6 or older than 12 years of age
* do not live within 2 miles of study park
* already meet physical activity guidelines
* not able to be physically active plan to move within two years

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 430 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Minutes per day of moderate and vigorous physical activity | two years
  Accelerometers worn for 7 day calculate minutes per day of moderate and vigorous physical activity
Minutes per day of light and sedentary activity | two years
  Accelerometers worn for 7 days calculate minutes per day of light and sedentary activity

CONTACTS AND LOCATIONS:
Overall Officials: Simone A French, PhD, Principal Investigator — University of Minneaots
Locations (1):
- University of Minnesota Division of Epidemiology & Community Health, Minneapolis, Minnesota, United States